CLINICAL TRIAL: NCT06953414
Title: Classification and Prediction of Difficult Awake Tracheal Intubation With Flexible Bronchoscopes
Acronym: AirWake
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-101447-BO-ff
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Airway Management; Intubation, Intratracheal; Bronchoscopy; Endoscopes
Keywords: Airway management; Classification; Flexible endoscopy guided intubation; Fibroptic guided intubation; Respiratory system; Laryngeal diseases; Health records
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Airway management problems are key drivers for anesthesia-related adverse events. Awake tracheal intubation using flexible bronchoscopes with preserved spontaneous breathing (ATI:FB) is a recommended technique to manage difficult tracheal intubation in anesthesia, intensive care and emergency medicine. However, a prospective developed classification for this type of airway management is lacking. Due to the absence of a specifically tailored, validated classification for awake intubation with flexible bronchoscopes, many airway operators and institutions use classification tools that were originally developed for direct laryngoscopy, such as the percentage of glottic opening (POGO) score or Cormack-Lehane classification, although their diagnostic performance for the classification of ATI:FB is unknown. This prospective model development and validation study aims to develop two multivariable prediction models: a diagnostic prediction model to classify difficult ATI:FB after ATI:FB has been performed and a second prognostic prediction model to predict the risk for difficult ATI:FB before ATI:FB is performed. An additional aim is to develop a machine learning algorithm to evaluate ATI:FB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an anticipated difficult airways scheduled for ATI:FB
* Consent by the patient
* Minimum 18 years of age

Exclusion Criteria:

* Patients not scheduled for ATI:FB
* Pregnant or breastfeeding patients
* Consent not given by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anticipated difficult airways scheduled for surgery with general anaesthesia and tracheal intubation at a single study center
Sampling Method: Probability Sample
Enrollment: 313 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Difficult awake flexible bronchoscopic intubation | 1 hour
  Difficult airway alert issued by the airway operator following ATI:FB

SECONDARY OUTCOMES:
First attempt success | 1 hour
  Number of participants with successful ATI:FB with only one attempt
Number of bronchoscopy attempts | 1 hour
  Observed during airway management
Number of intubation attempts | 1 hour
  Observed during airway management
Successful ATI:FB | 1 hour
  Number of participants with successful ATI:FB
Successful bronchoscopy | 1 hour
  Number of participants with successful bronchoscopy
Successful tube placement | 1 hour
  Number of participants with successful tracheal tube placement
Coversion to another type of airway management | 1 hour
  Observed during airway management
Conversion from transnasal to transoral bronchoscopy or vice versa | 1 hour
  Observed during airway management
Percentage of glottic opening | 1 hour
  Grading of the best view obtained during laryngoscopy (%)
Glottic view | 1 hour
  Grading of the best view obtained using landmarks (6-stages)
Time to best glottic view | 1 hour
  Recorded during airway management (seconds)
Time to intubation | 1 hour
  Recorded during airway management (seconds)
Lowest oxygen saturation | 1 hour
  Measured during airway management (%)
Endtidal CO2 | 1 hour
  First value measured after intubation (mmHg)
Airway obstructions requiring external manipulation | 1 hour
  Observed during airway management
Hypoxia | 1 hour
  Observed during airway management
Cardiovascular event requiring intervention (hypotension/bradycardia) | 1 hour
  Relevant hypotension or bradycardia observed during airway management
Cardiovascular event requiring intervention (hypertension, tachycardia) | 1 hour
  Relevant hypertension or tachycardia observed during airway management
Additional manouvers and adjuncts used | 1 hour
  Observed during airway management
Patient discomfort during ATI:FB | 1 hour
  Observed during airway management
Airway-related complications | 1 hour
  Observed during airway management
Anaesthesia alert card issued | 1 hour
  Anaesthesia alert card issued by the airway operator
Recommendation for future airway management | 1 hour
  Recommendation documented by the airway operator after airway management
Richmond agitation-sedation Scale | 1 hour
  Observed during airway management (scale form -4 to 5 points; lower values indicate deeper sedation)
Subjective rating of difficulty of sedation, topicalisation, bronchoscopy and tube placement | 1 hour
  Rating of the airway operator (visual analog scales [0-100]; lower values indicate better conditions)
Preparation time | 1 hour
  Recorded during airway management

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, FEAMS, Principal Investigator — University Medical Center Hamburg-Eppendorf: Universitatsklinikum Hamburg-Eppendorf; Vera Köhl, MD, Principal Investigator — University Medical Center Hamburg-Eppendorf: Universitatsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Dohrmann T, Gutsche N, Kramer R, Zeidler EM, Roher K, Wunsch VA, Dankert A, Krause L, Zollner C, Sasu PB, Petzoldt M. Prospective development and validation of a universal classification for paediatric videolaryngoscopic tracheal intubation: the PeDiAC score. Anaesthesia. 2024 Nov;79(11):1201-1211. doi: 10.1111/anae.16394. Epub 2024 Aug 7. PMID 39108225
- [Background] Barclay-Steuart A, Grosshennig HL, Sasu P, Wunsch VA, Stadlhofer R, Berger J, Stark M, Sehner S, Zollner C, Petzoldt M. Transnasal Videoendoscopy for Preoperative Airway Risk Stratification: Development and Validation of a Multivariable Risk Prediction Model. Anesth Analg. 2023 Jun 1;136(6):1164-1173. doi: 10.1213/ANE.0000000000006418. Epub 2023 Apr 19. PMID 37074950
- [Background] Kohse EK, Siebert HK, Sasu PB, Loock K, Dohrmann T, Breitfeld P, Barclay-Steuart A, Stark M, Sehner S, Zollner C, Petzoldt M. A model to predict difficult airway alerts after videolaryngoscopy in adults with anticipated difficult airways - the VIDIAC score. Anaesthesia. 2022 Oct;77(10):1089-1096. doi: 10.1111/anae.15841. Epub 2022 Aug 25. PMID 36006056